CLINICAL TRIAL: NCT03412812
Title: A Phase I Dose Escalation Trial of Five Fraction Stereotactic Radiation Therapy for Brain
Brief Title: A Dose Escalation Trial of Five Fraction Stereotactic Radiation Therapy for Brain Metastases
Acronym: RAD1705
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, John Fiveash, MD, Assistant Professor - Department of Radiation Oncology, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300001065
Record Dates: First submitted 2017-12-29; First posted 2018-01-26 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Brain Metastases
Keywords: Brain Metastases; Stereotactic Radiosurgery
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 2.1-4.0 cm diameter (Experimental): Patients will undergo dose escalated five fraction stereotactic radiosurgery for diagnosed brain metastases. Only single largest tumor will be treated with dose escalation. All other tumors (if present) will be treated with standard of care five fraction stereotactic radiosurgery. Starting dose level 7 Gy x 5 fractions
  Interventions: Radiation: 7 Gy; Radiation: 8 Gy; Radiation: 9 Gy
- 4.1-6.0 cm diameter (Experimental): Patients will undergo dose escalated five fraction stereotactic radiosurgery for diagnosed brain metastases. Only single largest tumor will be treated with dose escalation. All other tumors (if present) will be treated with standard of care five fraction stereotactic radiosurgery. Starting dose level 6 Gy x 5 fractions.
  Interventions: Radiation: 6 Gy; Radiation: 7 Gy; Radiation: 8 Gy

INTERVENTIONS:
Radiation: 6 Gy — As focal radiation techniques are utilized more frequently in the treatment of brain metastases, there is increasing need to accurately define the appropriate patient and tumor characteristics for focal therapy. Unfortunately, not all patients are good candidates for single fraction stereotactic radiosurgery (SRS) since large tumors and those in unfavorable locations have been associated with unacceptable rates of treatment-related toxicity. Five fraction stereotactic radiation has proven to be a more effective treatment for these patients that aren't good candidates.
  Arms: 4.1-6.0 cm diameter
Radiation: 7 Gy — As focal radiation techniques are utilized more frequently in the treatment of brain metastases, there is increasing need to accurately define the appropriate patient and tumor characteristics for focal therapy. Unfortunately, not all patients are good candidates for single fraction stereotactic radiosurgery (SRS) since large tumors and those in unfavorable locations have been associated with unacceptable rates of treatment-related toxicity. Five fraction stereotactic radiation has proven to be a more effective treatment for these patients that aren't good candidates.
Radiation: 8 Gy — As focal radiation techniques are utilized more frequently in the treatment of brain metastases, there is increasing need to accurately define the appropriate patient and tumor characteristics for focal therapy. Unfortunately, not all patients are good candidates for single fraction stereotactic radiosurgery (SRS) since large tumors and those in unfavorable locations have been associated with unacceptable rates of treatment-related toxicity. Five fraction stereotactic radiation has proven to be a more effective treatment for these patients that aren't good candidates.
Radiation: 9 Gy — As focal radiation techniques are utilized more frequently in the treatment of brain metastases, there is increasing need to accurately define the appropriate patient and tumor characteristics for focal therapy. Unfortunately, not all patients are good candidates for single fraction stereotactic radiosurgery (SRS) since large tumors and those in unfavorable locations have been associated with unacceptable rates of treatment-related toxicity. Five fraction stereotactic radiation has proven to be a more effective treatment for these patients that aren't good candidates.
  Arms: 2.1-4.0 cm diameter

SUMMARY:
This study looks at dose escalation for five fraction stereotactic radiotherapy for patients diagnosed with brain metastases with tumors 2.1-4.0 cm in diameter or 4.1-6.0 cm in diameter.

DETAILED DESCRIPTION:
This study looks at dose escalation treatment in patients diagnosed with brain metastases. Treatment involve five fraction stereotactic radiotherapy for patients with brain tumors 2.1-4.0 cm in diameter or 4.1-6.0 cm in diameter and dose escalation treatment is delivered only to the single largest tumor while all other tumors are treated with standard of care practices if they are present. A dose escalation schedule is proposed based on the monitoring of CNS toxicity and tumor size of the largest tumor, given it falls into the parameters set on diameter.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histologically confirmed malignancy.
* All patients must have imaging suggestive of one or more brain metastases.
* Karnofsky performance status (KPS) ≥ 60
* Age > 18 years
* Patients must provide written informed consent to participate in the study.
* Patients must have less than or equal to 10 brain metastases as identified on brain MRI.

Exclusion Criteria:

* History of surgical resection to the tumor of interest
* History of radiation to the tumor of interest
* History of previous whole brain irradiation
* Receipt of systemic therapy within one week of planned radiation treatment except for hormonal agents.
* Patient is unable to have MRI or MRI contrast.
* Inability to meet the appropriate normal tissue dose constraints secondary to tumor location should result in exclusion of the patient / tumor.
* Patients with a non-index tumor (second tumor) greater than 3 cm in diameter will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-07-30 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2025-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Fiveash, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Hazelrig-Salter Radiation Oncology Center, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.1-4.0 cm diameter; 4.1-6.0 cm diameter: Patients will undergo dose escalated five fraction stereotactic radiosurgery for diagnosed brain metastases. Only single largest tumor will be treated with dose escalation. All other tumors (if present) will be treated with standard of care five fraction stereotactic radiosurgery.
Period: Level 1
Arm/Group | 2.1-4.0 cm diameter | 4.1-6.0 cm diameter
Started | 12 | 1
Completed | 9 | 0
Not Completed | 3 | 1
Not completed — Death | 3 | 0
Not completed — Adverse Event | 0 | 1
Period: Level 2
Arm/Group | 2.1-4.0 cm diameter | 4.1-6.0 cm diameter
Started | 0 (There were no eligible patients therefore the study stopped prior to level 2.) | 0
Completed | 0 | 0
Not Completed | 0 | 0
Period: Level 3
Arm/Group | 2.1-4.0 cm diameter | 4.1-6.0 cm diameter
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 2.1-4.0 cm diameter level 2 and level 3 did no enroll any subjects. Dose level 2 did not enroll due to no eligible subjects.
  4.1-6.0 cm diameter level 1 had one subject enrolled and they experienced seizures at day 86, this was considered a dose limiting event and not subjects were enrolled in level 2 or level 3.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.1-4.0 cm diameter | 4.1-6.0 cm diameter | Total
Number analyzed (Participants) | 12 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 1 | 9
  >=65 years | 4 | 0 | 4
Age, Continuous [Mean (Full Range); unit: years] | 65 [49 to 68] | 65 [65 to 65] | 65 [49 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 5 | 0 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 3 | 0 | 3
  Race: White | 9 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 12 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Five Fraction Stereotactic Radiotherapy
Description: To determine the maximum tolerated dose of five fraction stereotactic radiotherapy for patients with either tumors 2.1-4.0 cm in diameter or 4.1-6.0 cm in diameter
Time Frame: 1-2 years
Measure: Number; unit: Gy
Groups:
- Dose Escalated 5 Fraction Stereotactic Radiosurgery - 2.1-4.0 cm: Patients will undergo dose escalated five fraction stereotactic radiosurgery for diagnosed brain metastases. Tumors must fall into one of two categories: 2.1-4.0cm diameter. Only single largest tumor will be treated with dose escalation. All other tumors (if present) will be treated with standard of care five fraction stereotactic radiosurgery.
  Dose Escalated Five Fraction Stereotactic Radiosurgery: As focal radiation techniques are utilized more frequently in the treatment of brain metastases, there is increasing need to accurately define the appropriate patient and tumor characteristics for focal therapy. Unfortunately, not all patients are good candidates for single fraction stereotactic radiosurgery (SRS) since large tumors and those in unfavorable locations have been associated with unacceptable rates of treatment-related toxicity. Five fraction stereotactic radiation has proven to be a more effective treatment for these patients that aren't good candidates.
- Dose Escalated 5 Fraction Stereotactic Radiosurgery - 4.1-6.0 cm: Patients will undergo dose escalated five fraction stereotactic radiosurgery for diagnosed brain metastases. Tumors must fall into one of two categories: 4.1-6.0cm diameter. Only single largest tumor will be treated with dose escalation. All other tumors (if present) will be treated with standard of care five fraction stereotactic radiosurgery.
  Dose Escalated Five Fraction Stereotactic Radiosurgery: As focal radiation techniques are utilized more frequently in the treatment of brain metastases, there is increasing need to accurately define the appropriate patient and tumor characteristics for focal therapy. Unfortunately, not all patients are good candidates for single fraction stereotactic radiosurgery (SRS) since large tumors and those in unfavorable locations have been associated with unacceptable rates of treatment-related toxicity. Five fraction stereotactic radiation has proven to be a more effective treatment for these patients that aren't good candidates.
Arm/Group | Dose Escalated 5 Fraction Stereotactic Radiosurgery - 2.1-4.0 cm | Dose Escalated 5 Fraction Stereotactic Radiosurgery - 4.1-6.0 cm
Number analyzed (Participants) | 12 | 1
Gy | 35 | 30

2. Secondary Outcome: Acute Toxicity of Five Fraction Stereotactic Radiotherapy Using Adverse Event Questionnaire
Description: To assess the acute toxicity of five fraction stereotactic radiotherapy for tumors 2-6 cm in diameter using the RAD 1705 Adverse Events Assessment. This assessment was created within our department and will be used specifically for this study.
Time Frame: 1-2 years
Reporting Status: Not Posted

3. Secondary Outcome: Late Toxicity of Five Fraction Stereotactic Radiotherapy Using Adverse Event Questionnaire
Description: To assess the late toxicity of five fraction stereotactic radiotherapy for tumors 2-6 cm in diameter using the RAD 1705 Adverse Events Assessment. This assessment was created within our department and will be used specifically for this study.
Time Frame: 1-2 years
Reporting Status: Not Posted

4. Secondary Outcome: Rate of Local Tumor Control With Five Fraction Stereotactic Radiotherapy Using Adverse Event Questionnaire
Description: To determine the rate of local tumor control with five fraction stereotactic radiotherapy for tumors 2-6 cm in diameter using the RAD 1705 Adverse Events Assessment. This assessment was created within our department and will be used specifically for this study.
Time Frame: 1-2 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Feasibility of Capturing Patient Reported Outcomes Electronically Using FACT-Br Questionnaire
Description: To assess the feasibility of capturing patient reported outcomes with the Functional Assessment of Cancer Therapy-Brain Questionnaire (FACT-Br) electronically in the Radiation Oncology clinic
Time Frame: 1-2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | 2.1-4.0 cm diameter | 4.1-6.0 cm diameter
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/1
Serious Adverse Events (participants affected / at risk) | 6/12 | 1/1
Other Adverse Events (participants affected / at risk) | 0/12 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.1-4.0 cm diameter (N=12) | 4.1-6.0 cm diameter (N=1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Cognitive Disability (General disorders) | 1 (1) | 0 (0)
Radiation Necrosis (Surgical and medical procedures) | 1 (1) | 0 (0)
Stroke (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT03412812/Prot_SAP_000.pdf